CLINICAL TRIAL: NCT01856647
Title: A Pilot Study to Characterize Adipose Tissue Leukocytes by Flow Cytometry and Microscopy in Lean, Obese and Psoriatic Subjects (Lean/Obese)
Brief Title: Pilot Study Characterizing Adipose Tissue Leukocytes by Flow Cytometry/Microscopy in Lean, Obese and Psoriatic Subjects
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: JUG-0799
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Psoriasis; Obesity
Keywords: Psoriasis; Obesity
MeSH Terms: conditions — Psoriasis; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fat Biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- lean (BMI≤ 24.9 Kg/m2): Adipose tissue biopsy (fat biopsy) in 9 lean (BMI≤ 24.9 Kg/m2)
  Interventions: Procedure: Adipose tissue biopsy (fat biopsy)
- obese (BMI= 30-40 Kg/m2): 9 obese (BMI= 30-40 Kg/m2)
  Interventions: Procedure: Adipose tissue biopsy (fat biopsy)
- psoriatic lean: 9 psoriatic lean
  Interventions: Procedure: Adipose tissue biopsy (fat biopsy)
- psoriatic obese: 9 psoriatic obese
  Interventions: Procedure: Adipose tissue biopsy (fat biopsy)

INTERVENTIONS:
Procedure: Adipose tissue biopsy (fat biopsy) — An adipose tissue biopsy will be performed after a 10-12 hour overnight fast. A small sample of fat tissue will be removed from the subject for gene expression analysis. A subcutaneous fat biopsy (~3 ml) will be obtained from the lower abdomen following local anesthesia.

SUMMARY:
Obesity is an insulin resistance-associated metabolic disorder which is a hallmark of and risk factor for type 2 diabetes and the metabolic syndrome, often linked to cardiovascular disease, certain cancers and inflammatory diseases.The phenotyping of subcutaneous adipose tissue (SAT) hematopoetic cells from obese subjects by flow cytometry, microscopy and gene expression will enable us to identify inflammation in this tissue and may help us to understand the causes and consequences of obesity in order to determine how these cells might be implicated in the initiation and/or progression of the aforementioned diseases.

DETAILED DESCRIPTION:
Obesity is an insulin resistance-associated metabolic disorder which is a hallmark of and risk factor for type 2 diabetes and the metabolic syndrome. It is also often linked to cardiovascular disease, certain cancers (e.g., colorectal, esophageal, endometrial, and ovarian), and inflammatory diseases (e.g., psoriasis, osteoarthritis,inflammatory bowel disease).The phenotyping of subcutaneous adipose tissue (SAT) hematopoetic cells from obese subjects by flow cytometry, microscopy and gene expression will enable us to identify inflammation in this tissue and may help us to understand the causes and consequences of obesity in order to determine how these cells might be implicated in the initiation and/or progression of the aforementioned diseases.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic lean cohort (BMI between 18-24.9 Kg/m2): moderate to severe plaque-type, at least 5% of BSA
* Psoriatic obese cohort (BMI between 30-40 Kg/m2): moderate to severe plaque-type, at least 5% of BSA
* Lean/non-psoriatic cohort: BMI between 18-24.9 Kg/m2
* Overweight/obese non-psoriatic cohort: BMI between 30-40 Kg/m2
* Subjects must be 18-65 years of age

Exclusion Criteria:

* Having received any systemic treatment for psoriasis within the last 30 days
* history of bleeding disorder
* weight loss of 10 pounds in the last four weeks
* current smoker
* Known diagnosis of any unrelated autoimmune disease or inflammatory disease ( i.e. lupus, atopic dermatitis, rheumatoid arthritis).
* Currently taking NSAIDS, aspirin, (if > once a week, stopped <30 days ago). Aspirin 81mg may be permitted if the Framingham Risk Score is < 10
* Having received any anti-inflammatory medication within the last 30 days
* Current use of any anti-coagulants
* LFTs > 2 x upper normal limits
* HIV infection
* Pregnant
* Less than 6 weeks post partum
* history of cardiovascular disease (MI, CHF, CVA)
* Any cancer diagnosis within the last 5 years
* Symptoms of acute illness such as upper respiratory infection, bronchitis, gastroenteritis, or fever within 3 days of Visit 1
* Any medical, psychological or social condition that, in the opinion of the Investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data
* ingestion of DHA or fish oil within last 90 days
* hypertension as defined as > 140 systolic and > 90 diastolic after 10 minutes of resting on 2 antihypertensives
* Use of statins within the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obesity and psoriasis are characterized by infiltration of inflammatory cells (leukocytes) in SAT and skin, respectively. We expect that SAT in obese psoriasis subjects will have infiltrating inflammatory leukocytes because of obesity, and that these infiltrating leukocytes might be different and/or increased in numbers by the pathology of psoriasis
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Biomarkers for phenotyping a new type of leukocyte | 5 years
  Biomarkers for phenotyping a new type of leukocyte

CONTACTS AND LOCATIONS:
Overall Officials: Juana Gonzalez, Principal Investigator — Rockefeller Univesrity
Locations (1):
- The Rockefeller University, New York, New York, United States